CLINICAL TRIAL: NCT06513754
Title: Investigating Changes in Responses to Controlled Effective Doses of Ozone at Different Exercise Intensities
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is not a clinical trial.
Sponsor: Michael Koehle (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor-Investigator, Michael Koehle, Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: O3ED
Record Dates: First submitted 2024-05-25; First posted 2024-07-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Ozone; Exercise Intensity
Keywords: Ozone; Exercise Intensity; Pulmonary Function; Ventilation; Dyspnea
MeSH Terms: conditions — Respiratory Aspiration; Dyspnea | interventions — Ozone

STUDY DESIGN:
Intervention Model Description: The study design to be employed for this study can be characterized as a double-blind cross over. ozone status (room air (<10 ppb ozone) and 170 ppb ozone), exercise intensity (moderate and heavy), sex, lung size, and time will be independent variables
Who Masked: Participant, Investigator
Masking Description: Both participants and investigator will be blinded to ozone status using nose clips
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ozone, High Intensity (Experimental): Participants will exercise for 45 minutes in the heavy intensity domain while exposed to 180 ppb ozone
  Interventions: Other: Ozone; Behavioral: Heavy Intensity
- Ozone, Moderate Intensity (Experimental): Participants will exercise for 75 minutes in the moderate intensity domain while exposed to 180 ppb ozone
  Interventions: Other: Ozone; Behavioral: Moderate Intensity
- Filtered Air, Heavy Intensity (Sham Comparator): Participants will exercise for 45 minutes in the heavy intensity domain while exposed to filtered air.
  Interventions: Behavioral: Heavy Intensity; Other: Filtered Air
- Filtered Air, Moderate Intensity (Sham Comparator): Participants will exercise for 75 minutes in the moderate intensity domain while exposed to filtered air
  Interventions: Behavioral: Moderate Intensity; Other: Filtered Air

INTERVENTIONS:
Other: Ozone — Ozone is a pollutant that forms as a result of nitrogen oxides or volatile organic compounds interacting with UV radiation. Ozone will be created via a generator in the lab
  Other Names: O3
  Arms: Ozone, High Intensity; Ozone, Moderate Intensity
Behavioral: Heavy Intensity — Heavy intensity exercise between the first and second ventilatory threshold for 45 minutes
  Arms: Filtered Air, Heavy Intensity; Ozone, High Intensity
Behavioral: Moderate Intensity — Moderate intensity exercise below the first ventilatory threshold for approximately 75 minutes
  Arms: Filtered Air, Moderate Intensity; Ozone, Moderate Intensity
Other: Filtered Air — Exposure to filtered air (<10 ppb ozone)
  Arms: Filtered Air, Heavy Intensity; Filtered Air, Moderate Intensity

SUMMARY:
The project will look to investigate whether exercise during ozone exposure performed for a shorter duration at a higher intensity is more harmful than exercise performed for a longer duration at a lighter intensity. To assess this, participants will perform these exercise conditions with and without ozone exposure and researchers will assess changes in lung function, subjective symptoms, and breathing mechanics to determine which is more harmful.

DETAILED DESCRIPTION:
Purpose and Hypothesis The purpose of the study is to investigate whether exercise performed at a higher intensity for a shorter duration during ozone exposure results in greater decrements in pulmonary function, subjective symptoms, and dyspnea than low intensity exercise performed for a longer duration. The researcher's hypothesize that high intensity exercise will result in worsened responses as a result of changes to breathing mechanics resulting in greater penetration of ozone into smaller airways of the lungs.

Justification Due to the growing incidence of wildfires, temperature increase with climate change and increased urbanization, more people are exposed to high levels of ozone despite standards set by international and national agencies. Despite health warnings, many choose to continue engaging in exercise during high ozone levels. Results from this study will better inform practitioners and exercisers how to engage in exercise during ozone conditions to minimize it's deleterious effects on health.

Research Design This is a double-blinded randomized cross over design with pre- and post-measures. Ozone status (room air and 180 parts per billion (PPB) ozone) and exercise intensity (moderate and heavy) are the independent variables each with two levels. Testing will take place over 5 laboratory visits separated by at least 7 days. During the first session, subjects will undergo body plethysmography, spirometry, and a Step-ramp-step test on a cycle ergometer to determine subject characteristics and exercise thresholds. During visits 2-5, participants will be randomized to 1 of 4 exercise conditions manipulating exercise intensity and ozone status. They will then be asked to exercise for a duration that incurs the same effective dose of ozone across conditions with ozone exposure. If the participant is exercising in a non-ozone condition, they will be asked to exercise for however long it would take to incur the same effective dose had they been exposed to 180 ppb of ozone during the exercise bout. During the exercise bout, participants will be asked to rate their subjective symptoms associated with ozone exposure, dyspnea, and RPE every 15 minutes. Once the exercise bout is complete, participants will immediately perform pulmonary function testing and will be asked to rate their subjective symptoms associated with ozone exposure, dyspnea, and RPE.

Statistical Analysis To analyze changes in pulmonary function, dyspnea, and subjective symptoms within exercise conditions a repeated measures ANOVA will be conducted. To analyze changes in these variables across conditions relative to ozone status, exercise intensity, sex, and lung size, a multivariate ANOVA will be conducted. To test for significance within and across conditions, a Tukey test will be performed. All data analysis will be conducted in R. The sample size employed for the study will be 18 (n = 9 male, n =9 female)

ELIGIBILITY:
Inclusion Criteria:

1. Currently training and/or competing in endurance sport
2. Maximal oxygen consumption (VO2max) greater than 60 ml/kg/min (males) or 50 ml/kg/min (females)
3. Between the ages of 18 and 50
4. Able to communicate sufficiently using the English language
5. Taking hormonal birth control (female participants only)

Exclusion Criteria:

1. History of smoking
2. Upper respiratory tract infection within the last 4 weeks
3. EIB, Asthma
4. Presence of any chronic respiratory disease
5. Current symptoms of, or current infection with COVID-19
6. Pregnant or suspected pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function | Measured before, during, and after exercise (before, 45th minute of exercise, immediately after, and every 30 minutes after for an hour)
  forced vital capacity, forced expiratory volume in 1 second, forced expiratory flow over the middle half of FVC.

SECONDARY OUTCOMES:
Rating of perceived exertion | Measured during and after exercise (every 15 minutes during, immediately after, and every 30 minutes after for an hour)
  How hard does the exercise feel rated on a scale of 6-20 with each increase representing an increase in perceived exertion while exercising
Sensations of Dyspnea | Measured before, during, after exercise (before, every 15 minutes during, immediately after, and every 30 minutes after for an hour)
  Sensations of breathlessness as measured by the multidimensional dyspnea profile. Increased scores represent worsened sensations or severities of dyspnea.
Subjective Symptoms | Measured before, during, after exercise (before, every 15 minutes during, immediately after, and every 30 minutes after for an hour)
  Subjective symptoms associated with ozone exposure using a questionnaire previously used by the Environmental Physiology Laboratory. This scale measures the presence and severity of eye, throat, lung irritation in response to ozone exposure. Higher scores indicate worsened symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koehle, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Environmental Physiology Laboratory, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No